CLINICAL TRIAL: NCT02717546
Title: Zimmer® MotionLoc® in Distal Tibia Fractures: An Observational Study
Brief Title: Zimmer® MotionLoc® in Distal Tibia Fractures
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CSE2014-08T
Record Dates: First submitted 2016-02-22; First posted 2016-03-23 (Estimated); Results first posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Distal Tibia Fractures
Keywords: Distal Tibia Fracture Screw

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group One: Distal Tibia Fracture repaired with Zimmer MotionLoc Screw
  Interventions: Device: Zimmer MotionLoc Screw

INTERVENTIONS:
Device: Zimmer MotionLoc Screw — Patients with distal tibia fractures (AO 43-A and C) requiring surgical intervention eligible for locked plating.

SUMMARY:
The objective of this observational prospective study is to systematically document the clinical outcomes of Zimmer MotionLoc Screws for Periarticular Locking Plate System applied to distal tibia fracture treatment and confirm safety and performance of the screws.

DETAILED DESCRIPTION:
Primary Endpoint:

* Radiographic & clinical fracture healing at 3 months post-surgery.

Secondary Endpoints:

* Complications
* Radiologic & clinical fracture healing at 6 weeks, 3, 6, and 12 months post-surgery.
* Callus size & distribution at 6 weeks, 3, 6, and 12 months post-surgery.

Radiologic fracture healing is defined as bridging of three of the four cortices as seen on x-ray/CT. Clinical healing will be assessed using the Function Index for Trauma (FIX-IT). The FIX-IT instrument quantifies clinical healing by assessing weight-bearing and fracture site pain on an ordinal scale. It has been initially validated in patients with tibia and femur fractures.

Callus size of the anterior, posterior, and medial aspect will be assessed for each time point using a validated and published computational method.

ELIGIBILITY:
Inclusion Criteria:

* With or without fibula fracture involvement (treated or not treated by osteosynthesis)
* Close or open fractures Gustilo type I
* Unilateral or bilateral fractures
* Patients who are capable of understanding the doctor's explanations, following his instructions and are able to participate in the follow-up program.
* Patients who give written consent to take part in the study by signing the "Patient Consent Form".

Exclusion Criteria:

* Delay of surgery for more than two weeks.
* Open fractures Gustilo type II & III
* History of infection of the affected extremity
* Non-ambulatory patients
* Planned fixation strategy includes interfragmentary lag screw fixation of non-articular fractures.
* Addition of bone graft, bone graft substitute or bone morphogenetic protein (BMP).
* Immobilization with plaster.
* Likely problems with maintaining follow-up program (e.g. patients with no fixed address, plans to move during course of study)
* Not expected to survive the duration of follow-up program.
* Patients known to be pregnant or breastfeeding.
* Patients who are unwilling or unable to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-02; Primary Completion 2019-12-05 (Actual); Study Completion 2020-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kacy Arnold, RN MBA, Study Director — Zimmer Biomet
Locations (7):
- United States (3):
  - Springfield Clinic, Springfield, Illinois
  - Indiana University, Indianapolis, Indiana
  - Donald B. Slocum Research and Education Foundation, Eugene, Oregon
- Mackay Specialist Day Hospital, Mount Pleasant, Australia
- Azienda Ospedaliera Universitaria Senese, Siena, Italy
- Korea University Anam Hospital, Seoul, South Korea
- The Dudley Group NHS Foundation Trust, Dudley, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group One
Started | 32
Completed | 20
Not Completed | 12
Not completed — Lost to Follow-up | 12

BASELINE CHARACTERISTICS:
Arm/Group | Group One
Number analyzed (Participants) | 32
Age, Continuous [Mean (Full Range); unit: years] | 53.5 [24 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 3
  United States | 12
  Italy | 13
  Australia | 4

OUTCOME MEASURES:

1. Primary Outcome: Average Clinical Fracture Healing of the Tibia Using the Function Index for Trauma (FIX-IT) Score at 3 Months Follow-up
Description: This measure will be assessed using the Function Index for Trauma (FIX-IT). The instrument quantifies clinical healing by assessing weight-bearing and fracture site pain on an ordinal scale. Minimum (worst) score possible is 0 and Maximum (best) score possible is 12.
Time Frame: 3 months
Population: Thirty-two subjects were enrolled globally. At 3 months follow-up, 29 subjects completed their visit and contributed to study data collection, thus 29 subjects were analyzed for this 3 month primary endpoint. However, the participation flow reports 20 subjects completed, which is reporting the number of subjects that were available for data collection at the 12 month follow-up.
Measure: Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Group One
Number analyzed (Participants) | 29
score on scale | 7.5 [6.6 to 8.4]

2. Primary Outcome: Number of Participants With Radiographic Fracture Healing of the Tibia at 3 Months Follow-up
Description: Radiographic fracture healing is defined as bridging of three of the four cortices (as seen on x-ray/CT).
Time Frame: 3 months
Population: Thirty-two subjects were enrolled globally. After 3 months follow-up, 29 subjects remained in the study for data collection, thus 29 subjects were analyzed for the primary endpoint. However, the participation flow reports 20 subjects completed, which is reporting the number of subjects that were available for data collection at the 12 month follow-up.
Measure: Number; unit: participants
Arm/Group | Group One
Number analyzed (Participants) | 29
participants | 3

3. Secondary Outcome: Complications
Description: Adverse Events were summed for all time points for the totality of the study. I.E. - complications reported for all sites at 6 weeks, 3 months, 6 months, and 12 months were summed and reported as a single secondary outcome measure for the study.
Time Frame: 12 months
Population: Complications were reported for all 32 subjects. If a subject was lost to follow-up, all existing complications for that subject remained in the data for reporting.
Measure: Number; unit: adverse events
Arm/Group | Group One
Number analyzed (Participants) | 32
adverse events
  Adverse Events | 8
  Device Related Adverse Events | 3

4. Secondary Outcome: Average Clinical Fracture Healing of the Tibia Using the Function Index for Trauma (FIX-IT) Score at 6 Weeks Follow-up
Description: This measure will be assessed using the Function Index for Trauma (FIX-IT) The instrument quantifies clinical healing by assessing weight-bearing and fracture site pain on an ordinal scale. Minimum (worst) score possible is 0 and Maximum (best) score possible is 12.
Time Frame: 6 weeks
Population: Thirty-two subjects were enrolled globally. At 6 weeks follow-up, 28 subjects completed their visit and contributed to study data collection, thus 28 subjects were analyzed for this 6 week secondary endpoint. However, the participation flow reports 20 subjects completed, which is reporting the number of subjects that were available for data collection at the 12 month follow-up.
Measure: Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Group One
Number analyzed (Participants) | 28
score on scale | 4.4 [3.6 to 5.1]

5. Secondary Outcome: Average Clinical Fracture Healing of the Tibia Using the Function Index for Trauma (FIX-IT) Score at 6 Months Follow-up
Description: as for outcome 4
Time Frame: 6 months
Population: Thirty-two subjects were enrolled globally. At 6 months follow-up, 27 subjects completed their visit and contributed to study data collection, thus 27 subjects were analyzed for this 6 month secondary endpoint. However, the participation flow reports 20 subjects completed, which is reporting the number of subjects that were available for data collection at the 12 month follow-up.
Measure: Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Group One
Number analyzed (Participants) | 27
score on scale | 10.9 [10.1 to 11.6]

6. Secondary Outcome: Average Clinical Fracture Healing of the Tibia Using the Function Index for Trauma (FIX-IT) Score at 12 Months Follow-up
Description: as for outcome 4
Time Frame: 12 months
Population: Thirty-two subjects were enrolled globally. At 12 months follow-up, 20 subjects completed their visit and contributed to study data collection, thus 20 subjects were analyzed for this 12 month secondary endpoint.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group One
Number analyzed (Participants) | 20
score on a scale | 11.5 [11 to 12]

7. Secondary Outcome: Number of Participants With Radiographic Fracture Healing of the Tibia at 6 Weeks Follow-up
Description: Radiographic fracture healing is defined as bridging of three of the four cortices (as seen on x-ray/CT).
Time Frame: 6 weeks
Population: Thirty-two subjects were enrolled globally. After 6 weeks follow-up, 28 subjects completed their visit and contributed to study data collection, thus 28 subjects were analyzed for this 6 week secondary endpoint. However, the participation flow reports 20 subjects completed, which is reporting the number of subjects that were available for data collection at the 12 month follow-up.
Measure: Number; unit: participants
Arm/Group | Group One
Number analyzed (Participants) | 28
participants | 2

8. Secondary Outcome: Number of Participants With Radiographic Fracture Healing of the Tibia at 6 Months Follow-up
Description: Radiographic fracture healing is defined as bridging of three of the four cortices (as seen on x-ray/CT).
Time Frame: 6 months
Population: Thirty-two subjects were enrolled globally. After 6 months follow-up, 27 subjects completed their visit and contributed to study data collection, thus 27 subjects were analyzed for this 6 month secondary endpoint. However, the participation flow reports 20 subjects completed, which is reporting the number of subjects that were available for data collection at the 12 month follow-up.
Measure: Number; unit: participants
Arm/Group | Group One
Number analyzed (Participants) | 27
participants | 14

9. Secondary Outcome: Number of Participants With Radiographic Fracture Healing of the Tibia at 12 Months Follow-up
Description: Radiographic fracture healing is defined as bridging of three of the four cortices without fracture line (as seen on x-ray/CT).
Time Frame: 12 months
Population: Radiographic fracture healing at 12 months follow-up for subjects that completed their clinic visit, or showed radiographic union prior to lost to follow-up. Twenty subjects completed their 12 month follow-up visit, of these, 15 showed radiographic union. In addition to these 15 subjects, 4 subjects had previously shown radiographic healing; however, they did not complete their 12 month protocol visit but were included in this 12 month results for a total of 24 participants analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Group One
Number analyzed (Participants) | 24
Participants | 19

ADVERSE EVENTS:
Time Frame: Per the protocol, ISO definitions were followed for adverse event data collection. All adverse events were captured for subjects enrolled through 12 months follow-up or study completion (including lost to follow-up), whichever came first.
Description: ISO definition is not materially different from clinicaltrials.gov definitions.
Arm/Group | Group One
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 1/32
Other Adverse Events (participants affected / at risk) | 6/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group One (N=32)
Compartment Syndrome (Vascular disorders) | 1 (32)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group One (N=32)
Patient diagnosed with diabetes. (Endocrine disorders) | 1
Evaluated for DVT (Swelling and pain). (Vascular disorders) | 1
Ankle collapse -9 degrees varus. (Product Issues) | 1
Evaluated for DVT. (Vascular disorders) | 1
Pop in operative leg followed by pain. (Product Issues) | 1
Painful hardware. (Product Issues) | 1
Left hip pain. (Musculoskeletal and connective tissue disorders) | 1
Scant serious drainage. (Infections and infestations) | 1
Diarrhea (Gastrointestinal disorders) | 1
Numbness in knee (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-30): https://cdn.clinicaltrials.gov/large-docs/46/NCT02717546/Prot_SAP_000.pdf